CLINICAL TRIAL: NCT03055663
Title: A Comparison of Patient Satisfaction Between Sedation Using Medication and Sedation Using Virtual Reality During Surgery Under Spinal Anesthesia: A Randomized Controlled Trial
Brief Title: Sedation Using Virtual Reality During Surgery Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1611-069-808
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Sedation; Spinal Anesthesia
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled trial
Masking Description: Open-labelled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality sedation (Experimental): Patients watches virtual reality sedation program that shows underwater world with comfortable music and narrations during surgery.
  Interventions: Other: Sedation by watching virtual reality sedative program
- Sedation with intravenous sedatives (Active Comparator): Patients receives intravenous sedative of midazolam (initial bolus 1-2 mg with maintenance dose of 1 mg every 10 - 30 min).
  Interventions: Procedure: Sedation by using intravenous sedative; Drug: Midazolam

INTERVENTIONS:
Other: Sedation by watching virtual reality sedative program — Patients watch three-dimensional virtual reality program with headset and headphone during surgery.
  Arms: Virtual reality sedation
Procedure: Sedation by using intravenous sedative — Patients receive intravenous sedative (midazolam 1-2 mg bolus with 1 mg maintenance dose every 10- 30 minutes)
  Arms: Sedation with intravenous sedatives
Drug: Midazolam — Patients receive intravenous sedative (midazolam 1-2 mg bolus with 1 mg maintenance dose every 10- 30 minutes)
  Arms: Sedation with intravenous sedatives

SUMMARY:
During spinal anesthesia, sedation is performed using intravenous sedative for the patient's comfort and appropriate surgical environment. However, side effects of medications such as respiratory depression, hypotension, bradycardia and desaturation cannot be avoided. Recently, there have been developed a virtual reality experience equipment and a variety of virtual reality programs including visuo-haptic computer technology. There have been clinical studies that apply this technology to the pain medicine, sedation and medical education. However, no study has been reported for the purpose of replacing sedation during spinal anesthesia.

Therefore, we attempt to evaluate the efficacy and safety of sedation using virtual reality meditation program during spinal anesthesia for urologic surgery.

DETAILED DESCRIPTION:
During spinal anesthesia, sedation is performed using intravenous sedative for the patient's comfort and appropriate surgical environment. However, side effects of medications such as respiratory depression, hypotension, bradycardia and desaturation cannot be avoided. Recently, there have been developed a virtual reality experience equipment and a variety of virtual reality programs including visuo-haptic computer technology. There have been clinical studies that apply this technology to the pain medicine, sedation and medical education. However, no study has been reported for the purpose of replacing sedation during spinal anesthesia.

Therefore, we attempt to evaluate the efficacy and safety of sedation using virtual reality meditation program during spinal anesthesia for urologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spinal anesthesia for urologic surgeries including Holmium Laser Enucleation of the Prostate or TransUrethral Resection of Bladder tumor).
* American Society of Anesthesiologists physical status classification 1, 2 or 3.
* Patients who voluntarily decides to participate in the trial and has given informed consent to this trial

Exclusion Criteria:

* History of chronic use of sedative, narcotics, alcohol or drug abuse
* Baseline oxygen saturation < 90%
* Baseline hemodynamic or respiratory instability (initial systolic blood pressure < 80 mmHg, respiratory rate > 25 breaths/min or < 10 breaths/min)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Satisfaction score of patient | 20 minutes after the arrival at the postanesthesia care unit
  Patient's satisfaction score measured by 5-point Likert-like verbal rating scale

SECONDARY OUTCOMES:
Satisfaction score of surgeon | 5 minutes after the end of the main surgical procedure
  Surgeon's satisfaction score measured by 5-point Likert-like verbal rating scale
Satisfaction score of anesthesiologist | 5 minutes after the end of the surgery
  Anesthesiologist's satisfaction score measured by 5-point Likert-like verbal rating scale
incidence of adequate sedation | 5 minutes after the end of surgery
  Adequate sedation is defined if all the following criteria met
  1. patient does not complain discomfort or does not move arm or face unnecessarily or intend to remove the monitoring device or cable
  2. patients lying still in a stable state
  3. incidence of desaturation (<95% for more than 5 sec) less than 2 (one or zero) during surgery
  4. incidence of apnea (duration of more than 5 seconds) less than 2 during surgery
  5. does not need mask ventilation or laryngeal mask insertion or endotracheal intubation
  6. incidence of hypotension (mean blood pressure<55 mmHg) or bradycardia (heart rate <50) less than 2 during surgery
  7. does not need propofol as a rescue sedative medication
incidence of desaturation | 5 min after the end of surgery
  incidence of desaturation (pulse oximetry <90% for more than 5 sec) during the surgery
incidence of apnea | 5 min after the end of surgery
  incidence of apnea (no detectable end-tidal carbon dioxide for more than 5 sec) during the surgery
incidence of hypotension | 5 min after the end of surgery
  incidence of hypotension (decrease in mean blood pressure of more than 30% of baseline or mean blood pressure less than 55 mmHg) during the surgery
incidence of bradycardia | 5 min after the end of surgery
  incidence of bradycardia (decrease in heart rate of more than 30% of baseline or heart rate fall below 50 beats/min
incidence of rescue medication for sedation | 5 min after the end of surgery
  incidence of rescue medication for sedation administered during the surgery
incidence of assisted mask ventilation | 5 min after the end of surgery
  incidence of assisted mask ventilation due to prolonged apnea during the surgery
incidence of nausea | 5 min after the end of surgery
  incidence of nausea of numerical rating scale of more than 5 during the surgery
incidence of vomiting | 5 min after the end of surgery
  incidence of vomiting during the surgery
time to recovery at post-anesthesia care unit | 5 min after the stay in the post-anesthesia care unit
  time to report the modified Aldrete score of 9 or more at post-anesthesia care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No